CLINICAL TRIAL: NCT06613464
Title: The Impact of Point-of-care Ultrasound on Treatment Planning and Prognosis in the Intensive Care Unit
Brief Title: The Impact of POCUS on Treatment Planning and Prognosis in the ICU
Status: Completed | Type: Observational
Sponsor: Döndü Genc Moralar (Other Government)
Responsible Party: Sponsor-Investigator, Döndü Genc Moralar, Assoc. Prof., Gaziosmanpasa Research and Education Hospital
Organization: Gaziosmanpasa Research and Education Hospital (Other Government)
Other Study IDs: 88
Record Dates: First submitted 2024-09-20; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: All of the Icu Patients Over 18 Years Old Except Pregnant, Trauma and AKI Patients
Keywords: POCUS; Ultrasound; Mortality
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ICU patients: Patients over the age of 18 who are admitted to intensive care unit and who have been in intensive care for >5 days
  Interventions: Diagnostic Test: diagnosis confirmation

INTERVENTIONS:
Diagnostic Test: diagnosis confirmation — The patients diagnoses will be confirmed though imaging methods like computed tomography chest x-ray and anamnesis

SUMMARY:
This study aims to understand how using bedside ultrasound in the intensive care unit (ICU) can improve diagnosis and treatment for critically ill patients. When patients are admitted to the ICU, doctors usually rely on various tests and assessments, such as the APACHE-II score, to estimate the severity of their condition and predict their chances of survival. In addition to these tests, we will use bedside ultrasound to examine the lungs, heart, vena cava (a large vein), and optic nerve, which can give us important information about the patient's condition.

By using ultrasound, we can look for things like fluid in the lungs, heart function, or increased pressure in the brain. Based on what we find with the ultrasound, we may adjust treatments, such as changing the amount of fluids given or starting new medications.

We will also compare each patient's condition on the first day and the fifth day, using both ultrasound findings and their APACHE-II score, to see if the ultrasound results have influenced their care and outcomes. The study will include 40 patients, and we will track their progress, including how long they stay on mechanical ventilation, how long they are in the hospital, and their survival after 28 days.

This research will help us learn more about how ultrasound can help doctors make better decisions in the ICU, leading to improved care for critically ill patients.

DETAILED DESCRIPTION:
### Detailed Description for Clinical Trials

This prospective observational study focuses on the routine use of point-of-care ultrasound (POCUS) in the intensive care unit (ICU) and its impact on diagnosis, treatment decisions, and patient outcomes. Bedside ultrasound is increasingly recommended in ICU settings because it provides non-invasive, repeatable, and immediate diagnostic information that can guide the management of critically ill patients.

Upon admission, all ICU patients will undergo an initial assessment, including routine tests such as the APACHE-II score, which helps to estimate the severity of illness and predict the likelihood of survival. The goal of this study is to evaluate how POCUS, in addition to standard care, influences patient outcomes and whether it provides any additional diagnostic information that changes the treatment plan.

Key components of the study include:

1. **Initial Evaluation:**

   * All patients will have their medical history taken, undergo a physical examination, and have blood tests performed, which are standard for ICU patients. These will be used to calculate the APACHE-II score.
   * In addition to routine care, each patient will be evaluated with POCUS, including:
   * **Lung Ultrasound (LUS):** The lungs will be divided into six regions (upper and lower parts of the anterior, lateral, and posterolateral thoracic walls) to check for conditions such as lung consolidation, edema, pleural effusion, or pneumothorax.
   * **Cardiac Ultrasound:** The heart will be examined for valvular pathologies, fractional shortening (FS), pericardial effusion, and inferior vena cava (IVC) diameter to assess volume status using the collapsibility and distensibility index.
   * **Optic Nerve Ultrasound:** The optic nerve sheath diameter will be measured to evaluate intracranial pressure.
2. **Changes in Diagnosis and Treatment:**

   * Based on the findings from the ultrasound, the treatment plan may be modified. For example, if the ultrasound reveals fluid overload or inadequate volume, the amount of intravenous fluids may be adjusted. If lung ultrasound shows consolidations, adjustments to patient positioning or additional interventions may be made. Similarly, changes in cardiac ultrasound may result in modifying inotropic or vasodilator therapy, and optic nerve measurements may influence treatments for brain edema.
   * After 5 days, the patients will undergo another ultrasound, and their APACHE-II score will be recalculated to assess the effectiveness of the treatments and any changes in patient prognosis.
3. **Outcome Measurement:**

   * The study will follow 40 patients over a 28-day period. Outcomes will be evaluated by comparing the initial and subsequent ultrasound findings, changes in treatment, and the predicted mortality rates based on the APACHE-II score.
   * Secondary outcomes will include the duration of mechanical ventilation, length of ICU stay, and 28-day mortality.
   * The study will also assess the impact of ultrasound on specific organ systems:
   * **Respiratory System:** LUS, PaO2/FiO2 ratio, and PaCO2 levels will be monitored to assess lung function.
   * **Cardiovascular System:** Intravascular volume will be evaluated using vena cava ultrasound, while heart failure will be assessed with FS and LUS scores.
   * **Intracranial Pressure:** The optic nerve sheath diameter will be used to monitor changes in intracranial pressure.

The primary objective of this study is to determine whether bedside ultrasound can provide additional diagnostic information that significantly impacts treatment decisions and improves patient outcomes in the ICU. The secondary aim is to evaluate the effect of ultrasound on the functionality of different organ systems and how it contributes to overall patient prognosis and survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who are admitted to intensive care
* Patients who have been in intensive care for more than 5 days

Exclusion Criteria:

* Being pregnant
* Patients with head trauma
* Acute renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to intensive care over the age of 18 and who have been in intensive care for more than 5 days
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
POCUS effectiveness | First 5 days
  The primary goal of our study is to evaluate the effectiveness of point-of-care ultrasound (POCUS) in the diagnosis and treatment of patients admitted to the intensive care unit (ICU). We aim to investigate how the use of ultrasound alters diagnostic clarity and treatment interventions compared to initial diagnoses made without ultrasound. Any new or additional diagnoses made following ultrasound will be considered supplemental findings, which may lead to changes in the treatment plan.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pontet J, Yic C, Diaz-Gomez JL, Rodriguez P, Sviridenko I, Mendez D, Noveri S, Soca A, Cancela M. Impact of an ultrasound-driven diagnostic protocol at early intensive-care stay: a randomized-controlled trial. Ultrasound J. 2019 Sep 30;11(1):24. doi: 10.1186/s13089-019-0139-2. PMID 31595353
- [Background] Manno E, Navarra M, Faccio L, Motevallian M, Bertolaccini L, Mfochive A, Pesce M, Evangelista A. Deep impact of ultrasound in the intensive care unit: the "ICU-sound" protocol. Anesthesiology. 2012 Oct;117(4):801-9. doi: 10.1097/ALN.0b013e318264c621. PMID 22990179